CLINICAL TRIAL: NCT06287320
Title: The Peripheral Blood Lymphocyte Subsets as Predicative Biomarkers Reflecting the Efficacy and Toxicity in Patients With Locally Advanced Non-small Cell Lung Cancer Received Chemoradiotherapy With or Without Immunotherapy
Brief Title: The Predictive Biomarkers in Patients With Locally Advanced Non-small Cell Lung Cancer
Status: Recruiting | Type: Observational
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: Bioplc
Record Dates: First submitted 2024-02-23; First posted 2024-03-01 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-01

CONDITIONS: Locally Advanced Non-small Cell Lung Cancer
Keywords: Peripheral blood lymphocyte subsets
MeSH Terms: interventions — Immunotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 10 ml whole blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- NSCLC patients received CRT plus ICIs: For it's an observational study, locally advanced NSCLC patients received CRT with induction immunotherapy or consolidation immunotherapy will be divided into the group "NSCLC patients received CRT plus ICIs".
  Interventions: Radiation: concurrent or sequential chemoradiotherapy; Drug: Immunotherapy
- NSCLC patients received CRT: For it's an observational study, locally advanced NSCLC patients received CRT without immunotherapy will be divided into the group "NSCLC patients received CRT".
  Interventions: Radiation: concurrent or sequential chemoradiotherapy

INTERVENTIONS:
Radiation: concurrent or sequential chemoradiotherapy — Thoracic radiation therapy(with the prescribed dose of 50-70 Gy), concurrently or sequentially combined with platinum-based doublet chemotherapy.
Drug: Immunotherapy — anti-PD-1/anti-PD-L1 immune checkpoint inhibitors
  Groups: NSCLC patients received CRT plus ICIs

SUMMARY:
This study is a prospective cohort study to evaluate the peripheral blood lymphocyte subsets as predicative biomarkers reflecting the efficacy and toxicity in patients with locally advanced non-small cell lung cancer (NSCLC) received chemoradiotherapy (CRT) with or without immune checkpoint inhibitors (ICIs).

DETAILED DESCRIPTION:
All patients had a pathologically confirmed locally advanced NSCLC according to the 8th AJCC staging system and received definitive radiotherapy, concurrently or sequentially combined with platinum-based doublet chemotherapy. The peripheral blood samples at various time points including before radiation, 4 weeks after beginning of radiation, the end of radiation, 1 month post radiation, and 1 month post consolidation immunotherapy were collected for lymphocyte subsets detection.

The subjects will be divided into two groups according to whether patients received ICIs, namely, NSCLC patients received CRT plus ICIs and NSCLC patients received CRT.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years; ECOG score 0-2.
2. Pathologically confirmed locally advanced NSCLC according to the 8th AJCC staging system.
3. Received definitive radiotherapy, concurrently or sequentially combined with platinum-based doublet chemotherapy.
4. No serious medical diseases and dysfunction of major organs, such as blood routine, liver, kidney, heart and lung function.

Exclusion Criteria:

1. Pathologic type was adenocarcinoma with EGFR gene mutation or ALK gene rearrangement.
2. Patients with other active malignancies within 5 years or at the same time.
3. Active or previously documented autoimmune or inflammatory diseases (including inflammatory bowel disease, diverticulitis [except diverticular disease], systemic lupus erythematosus, Sarcoidosis syndrome, Wegener' s syndrome).
4. History of allogeneic organ transplantation.
5. History of active primary immunodeficiency.
6. Patients with uncontrolled concurrent diseases, including but not limited to persistent or active infection (including tuberculosis, hepatitis B, hepatitis C, human immunodeficiency virus, etc.), symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, uncontrolled arrhythmia, active interstitial lung disease, severe chronic gastrointestinal disease with diarrhea or mental illness.
7. Women of child-bearing potential who are pregnant or breastfeeding.
8. The investigator judged other situations not suitable for inclusion in this study.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Consecutive locally advanced NSCLC patients treated with definitive CRT with or without ICIs at hospital.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Adverse Event | AEs and SAEs must be collected from the start of treatment to 28 days after discontinuation of study drug, up to 24 months.
  The incidence of adverse events (AEs) and serious adverse events (SAEs) is evaluated by CTCAE 5.0. Appropriate description of AEs and laboratory data/vital signs will be produced. Number of patients who had at least one adverse event will be calculated.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | From date of first treatment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months.
  Defined as the time from date of first treatment until the date of first documented progression or date of death from any cause, whichever came first.
Overall survival (OS) | From the date of first treatment to the date of any documented death due to any cause, assessed up to 24 months.
  Defined as the time from the date of first treatment to the date of any documented death due to any cause.
Objective Response Rate (ORR) | Tumor assessment using RECIST will be performed at baseline then every 3 months from the first treatment until objective progression or death from any cause, assessed up to 24 months.
  The objective response rate (ORR) will be calculated as the number of patients with CR or PR per RECIST Criteria.
  Complete Response (CR): Disappearance of all target lesions; Partial Response (PR): >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Disease control rate (DCR) | Tumour assessment using RECIST will be performed at baseline then every 3 months from first treatment until objective progression or death from any cause, assessed up to 24 months.
  DCR will be calculated as the number of patients with CR, PR or sustained SD≥6 weeks per RECIST Criteria.
  Complete Response (CR): Disappearance of all target lesions; Partial Response (PR): >=30% decrease in the sum of the longest diameter of target lesions; Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase.

CONTACTS AND LOCATIONS:
Overall Officials: Nan Bi, MD, Principal Investigator — Chinese Academy of Medical Sciences and Peking Union Medical College
Locations (1):
- Chinese Academy of Medical Science and Peking Union Medical College, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No